CLINICAL TRIAL: NCT03164122
Title: EVALUATION OF AN INNOVATIVE TREATMENT FOR RADIOCARPAL OSTEOARTHRITIS USING INTRA-ARTICULAR INJECTION OF A MIXTURE OF AUTOLOGOUS MICROFAT AND AUTOLOGOUS PLATELET-RICH PLASMA
Acronym: AMIPREP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-34; 2016-002648-18 (EudraCT Number)
Record Dates: First submitted 2017-05-19; First posted 2017-05-23 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intra-articular injection (Experimental)
  Interventions: Drug: injection of microfat and plasma rich platelet PRP; Device: MRI

INTERVENTIONS:
Drug: injection of microfat and plasma rich platelet PRP — intra-articular injections
Device: MRI — MRI 3T

SUMMARY:
Recently, the emergence of biotherapies has allowed the use of intra-articular injections of autologous plasma rich platelet (PRP). Their use is widespread since 2010 and is based on the demonstration that platelets-enriched plasma, by virtue of its growth factors concentration, stimulates in vitro and in vivo cartilage regeneration in preclinical models. Recent literature highlights that these autologous products are very well tolerated by humans. PRP, as an intra-articular injection therapy, seems to be an autologous biological medicine, innovative for cartilage injury reparation and showing good primary results for this indication.

Adipose tissue contains stromal-vascular fraction (SVF), in which are located a large proportion of mesenchymal multipotent stem cells (Adipose-derived stem cells, ADSCs) able to differentiate into several cellular lines in vitro and in vivo, including cartilage cells.

The association of microfat and PRP is interesting in order to potentiate trophic and regenerative effects on damaged cartilage site. The combination of these two products, respectively rich in autologous multipotent stem cells and growth factors, aims to create an optimal environment for cartilage cells regeneration. Furthermore, microfat semi solid phase is playing the role of a nutritive support matrix which contains and limits the diffusion and resorption of PRP liquid while allowing progressive growth factors release on the injection site.

The hypothesis of this project is that standardized injection of an innovative treatment (microfat and autologous PRP) should allow delay the use of invasive surgical therapy in the treatment of wrist osteoarthritis. This minimally invasive treatment could provide a curative second line treatment in case of medical treatment failure.

DETAILED DESCRIPTION:
Material and methods:

This research protocol aims to evaluate the safety of intra-articular injection of a mixture of autologous microfat associated with autologous PRP for radiocarpal osteoarthritis resistant to medical treatment.

This is a prospective, longitudinal, intrasubject, single-center clinical trial phase I-IIa evaluating the safety and feasibility of this innovative treatment.

Twelve patients will receive an intra-articular injection of 4 ml of an homogeneous mixture of autologous PRP (2ml) and microfat (2ml).

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 20 and 75 years of age
* Symptomatic radio-carpal osteoarthritis diagnosed by arthroscanner resistant to medical treatment and candidate to surgery
* BMI ≥ 20 Kg/m²
* Written informed consent, signed by patient or legal representative (if patient unable to sign).
* HB > 10g/dl
* Negative pregnancy test and efficiency contraception

Exclusion Criteria:

* - Thrombocytopenia < 150 G/L, Thrombocytosis > 450 G/L, Thrombopathy
* TP < 70%, TCA patient / witness rapport > 1,20
* Anemia: HB < 10g/dl
* Positive serology VIH1 and 2, Agp24, Ac HCV, Ag HbS, AcHbc, Ac HTLV I and II, TPHA
* Treatment by platelet inhibiting agent, aspirin, antivitamin K completed more than 2 weeks before inclusion
* Chronic treatment by corticosteroid per os or treatment completed more than 2 weeks before inclusion
* Intra articular injection of corticosteroid or hyaluronic acid completed more than 8 weeks before inclusion
* NSAI treatment completed more than 2 weeks before inclusion
* Fever or recent disease completed more than 1 month before inclusion
* Auto immune disease, Inflammatory or microcrystalline Arthritis, Immune deficit
* Infectious disease
* MRI contraindication: ocular loose bodies, pace maker, neurostimulator, cochlear implant, vascular clips, metallic cardiac val
* Anesthesia or surgery contra indication, iodine allergy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
evaluate the safety | 1 MONTH
  By the number of Adverse event related to the traitment

SECONDARY OUTCOMES:
Improvement of pain | 3 ,6, 12 months
  with the Visual Analogue Scale (VAS).
Improvement of wrist pain | 3 ,6, 12 months
  with DASH scores
Improvement of wrist pain and function | 3, 6,12 months
  with PWRE scores
Improvement of radiocarpal chondral lesions | 12 Months
  MRI

CONTACTS AND LOCATIONS:
Overall Officials: jean-olivier ARNAUD, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assisatnce Publique Hopitaux de Marseille, Marseille, France